CLINICAL TRIAL: NCT03625713
Title: Epidemiological, Clinical, Microbiological and Therapeutic Aspects of Sexually Transmitted Bacterial Ano-rectitis in a Specialized Consultation Center
Brief Title: Bacterial Ano-rectitis Sexually Transmitted in a Specialized Consultation Center
Acronym: IST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IST
Record Dates: First submitted 2018-07-13; First posted 2018-08-10 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Ano-Rectal Infection Bacterial Nos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infectious ano-rectitis is poorly described. Their epidemiology is poorly known, as are their clinical, diagnostic (diagnoses are regularly corrected in gastroenterology and new diagnostic tools are now available) and therapeutic aspects.

Analysis of data from this large population of patients referred to the proctology center for suspicion of Neisseria gonorrhoeae and / or Chlamydia trachomatis ano-rectitis will help identify risk factors and target prevention strategies and optimized therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Patient over the age of 18
* Patient consulting or hospitalized in the proctology center
* Patient for whom an anorectal sampling will be performed for suspicion of sexually transmitted infectious ano-rectitis

Exclusion Criteria:

* Patient's opposition to participate
* Patient deprived of liberty
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population corresponds to patients seen in hospital, in emergency consultation or programmed for a suspicion of infectious ano-rectitis and for whom a sampling for diagnostic purposes will be carried out and addressed in microbiology.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2024-06-02 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the clinical presentation | Day 1
  Prevalence of clinical signs : fever (yes/no), ulcerations (yes/no), purulent proctisis (yes/no), erythematosus proctisis (yes/no), condyloma (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent De Parades, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

IPD SHARING:
Plan to Share IPD: No